CLINICAL TRIAL: NCT00324961
Title: A 2-year Multi-centre, Open-label, Local Phase IV Study to Demonstrate the Efficacy and Safety of Adefovir Dipivoxil Tablets (10mg) in Chinese Subjects With HBe Antigen Negative Chronic Hepatitis B
Brief Title: Adefovir Dipivoxil Tablets (10mg) In Chinese Subjects With HBe Antigen Negative Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADF106632
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Results first posted 2009-10-02 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Chronic Hepatitis B
Keywords: adefovir dipivoxil; e Antigen negative; chronic hepatitis B; Chinese
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — adefovir dipivoxil

ARMS (1):
- Single arm open label adefovir dipivoxil (Experimental): adefovir dipivoxil once daily 10 mg orally
  Interventions: Drug: adefovir dipivoxil tablets

INTERVENTIONS:
Drug: adefovir dipivoxil tablets — adefovir dipivoxil once daily 10 mg orally

SUMMARY:
This is a phase IV, 2-year, multi-center, single arm and open-label study, evaluating the efficacy and safety with using local manufactured adefovir dipivoxil in Chinese subjects with HBeAg negative chronic hepatitis B

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-65 years inclusive
* Documented chronic hepatitis B infection determined by the presence of serum HBsAg for at least 6 months
* Documented HBeAg negative and HBeAb positive at the screening visit and with at least a 6 months history of HBeAg negativity.
* Serum HBV DNA ≥ 104 copies/mL (Roche COBAS AMPLICORTM HBV MONITOR Test, LLOD 300 copies/mL) at study screening (within 4 weeks before baseline)
* ALT value ≥1.3 times the upper limit of normal (ULN) at the time of screening, as determined using laboratory ranges and documented ALT abnormal within 6 month prior to the study screening.
* Serum alpha fetoprotein (AFP) < 50 ng/mL at the first screening visit. If the AFP level is ≥ 50 ng/mL but declined to < 50 ng/mL between screening and baseline, the patient is eligible.
* Compensated liver disease with the following laboratory and clinical parameters at study screening:

  * Prothrombin time ≤ 2 second above normal range.
  * Albumin ≥ 35 g/L.
  * Total bilirubin ≤ 2.5 mg/dL (≤ 43 µmol/L) or normal direct bilirubin.
  * No history of variceal bleeding.
  * No history of encephalopathy.
  * No history of ascites
  * Adequate renal function defined as serum creatinine ≤ 1.5 mg/dL (≤ 130 µmol/L).
  * Adequate hematological function defined as:
  * Absolute neutrophil count ≥ 1 x 10³/mm³ ( ≥ 1 x 10^9/L);
  * Platelets ≥ 80 x 10³/mm³ (≥ 80 x 10^9/L); Platelets ≥ 100 x 10³/mm³ ( ≥ 100 x 10^9/L) recommended for the patients who will undergo liver biopsy.
  * Hemoglobin ≥ 10 g/dL (≥ 100 g/L) (males) or ≥ 9 g/dL (≥ 9 g/L) (females).
  * Willing and able to undergo a minimum of two liver biopsies (prior to dosing, and after 104 weeks of therapy; only apply to subjects who are enrolled to the sites where liver biopsy is required).
  * A female is eligible to enter and participate in this study if she is of:

    1. non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is pre-menarchal or post-menopausal);
    2. child-bearing potential with a negative serum pregnancy test at screen, and agrees to one of the following: Complete abstinence from intercourse from 2 weeks prior to administration of the study drug, throughout the study, and for a time interval after completion or premature discontinuation from the study to account for elimination of the investigational drug, (a minimum of 5 half-lives or longer if the pharmacodynamic profile of the investigational drug warrants a longer time period); or, Female sterilization; or, Sterilization of male partner; or, Implants of levonorgestrel; or, Injectable progestogen; or, Oral contraceptive (combined or progestogen only); or, Any intrauterine device (IUD) with published data showing that the lowest expected failure rate is less than 1% per year (not all IUDs meet this criterion); or, Any other methods with published data showing that the lowest expected failure rate for that method is less than 1% per year; or, Barrier method only if used in combination with any of the above acceptable methods.
  * Agree not to participate in any other investigational trials or to undertake other HBV systemic antiviral regimens during participation in this study
  * Able to give written informed consent and comply with the requirements of the study

Exclusion Criteria:

* Any serious or active medical or psychiatric illnesses other than hepatitis B which, in the opinion of the investigator, would interfere with patient treatment, assessment or compliance with the protocol. This would include, may not limit to, renal, cardiac, pulmonary, vascular, neurogenic, digestive, metabolic (diabetes, thyroid disorders, adrenal disease), immunodeficiency disorders, active infection or cancer.
* Documented evidence of active liver disease due to other causes including co-infection hepatitis C (HCV), Subjects who are anti-HCV positive and in whom HCV RNA is undetectable are considered to be HCV seropositive and will not eligible; co-infection with hepatitis delta (HDV); co-infection with HIV; autoimmune hepatitis (antinuclear antibody titre > 1:160)
* Clinical signs of decompensated liver disease at baseline. These may include but are not limited to:

serum bilirubin > 2.5 mg/dL (≤ 43 µmol/L) - prothrombin time > 2 second prolonged above ULN

* serum albumin < 35g/L
* history of ascites, variceal bleeding, or encephalopathy

  * Alanine aminotransferase (ALT) >10 times ULN at screening or history of acute exacerbation leading to transient decompensation
  * Hepatocellular carcinoma as evidenced by one of the following:
* suspicious foci on ultrasound or radiological examination
* - where no positive ultrasound finding, but serum alpha-fetoprotein > 100ng/mL

  * Active alcohol or drug abuse or history of alcohol or drug abuse considered by the investigator to be sufficient to hinder compliance with treatment, participation in the study or interpretation of results.
  * Use of immunosuppressive therapy, immunomodulatory therapy (including interferon or thymosin), systemic cytotoxic agents, chronic anti-viral agents excluding lamivudine (e.g. ganciclovir, adefovir dipivoxil, entecavir, famciclovir, FTC, DAPD, LFMAU, HBIg), Chinese herbal medicines known to have activity against HBV within the previous 12 months or during the study; use of agents with effect of ALT reduction (e.g. schisandra agents) during the study
  * Use of lamivudine within the previous 3 months or during the study
  * Planned for liver transplantation or previous liver transplantation
  * Received hepatotoxic drugs (e.g., anabolic steroids, ketaconazole, itraconazole, isoniazid, rifampin, rifabutin) within 2 months prior to study screening or expected to receive these during the course of the study.
  * Received nephrotoxic drugs (e.g., aminoglycosides, amphotericin B, vancomycin, cidofovir, foscarnet, cis-platinum, pentamidine etc.) or competitors of renal excretion (e.g., probenecid) within 2 months prior to study screening or the expectation that patient will receive any of these during the course of the study.
  * Receiving systemic (intravenous or oral) steroids, immuno-suppressant therapies or chemotherapeutic agents within 2 months of study screening or expected to receive these agents during the course of the study.
  * History of hypersensitivity to nucleoside and/or nucleotide analogues.
  * Inability to comply with study requirements.
  * Lactating females or females with a positive serum pregnancy test.
  * Organ or bone marrow transplant recipients.
  * Previous (or planned) participation in an investigational trial involving administration of investigational compound within 2 months prior to the study screening.
  * Can not comply with the requirements of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 533 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- China (11):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Chongquin
  - GSK Investigational Site, Jinan
  - GSK Investigational Site, Shanghai

RESULTS

PARTICIPANT FLOW:
Groups:
- 10 mg Adefovir Dipivoxil (ADV): 10 mg ADV tablets once daily for 104 weeks
Period: Overall Study
Arm/Group | 10 mg Adefovir Dipivoxil (ADV)
Started | 533
Completed | 490
Not Completed | 43
Not completed — Adverse Event | 5
Not completed — Consent Withdrawn | 11
Not completed — Lost to Follow-up | 22
Not completed — Protocol Violation | 3
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | 10 mg Adefovir Dipivoxil (ADV)
Number analyzed (Participants) | 533
Age Continuous [Mean (Standard Deviation); unit: years] | 38.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121
  Male | 412
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 533

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving HBV DNA ≤300 Copies/mL at Week 104
Description: Hepatitis B Virus (HBV) DNA level is tested in blood serum by real-time Polymerase Chain Reaction with the lower limit of detection (LLD) as 300 copies/milliliter in a central laboratory.
Time Frame: Week 104
Population: Intent-to-Treat (ITT) Population: all HBeAg participants who actually received the study medication at least once. Participants with missing data were not included in the analysis.
Measure: Number; unit: participants
Groups:
- HBeAg- at Baseline: All participants who were Hepatitis B e Antigen (HBeAg) negative at baseline
Arm/Group | HBeAg- at Baseline
Number analyzed (Participants) | 488
participants
  HBV DNA ≤300 cp/mL | 85
  HBV DNA > 300 cp/mL | 403

2. Secondary Outcome: Number of Participants Achieving Histological Improvement After the 104-week Treatment
Description: Histological improvement (defined as ≥2 point reduction in the Knodell necroinflammation score without worsening fibrosis) was assessed by 2 independent pathologists in the HBeAg-negative participants who underwent 2 sequential liver biopsies at baseline and week 104/withdrawal. The Knodell/histological activity index (HAI) scoring system represents the sum of scores for periportal, bridging necrosis (0-10: none=0, multilobular necrosis=10), interlobular degeneration and focal necrosis (0-4: none=0, marked=4), portal inflammation (0-4: none=0, marked=4), and fibrosis (0-4: none=0, cirrhosis=4)
Time Frame: Week 104
Population: HBeAg negative chronic hepatitis B participants who underwent liver biopsy at Week 104
Measure: Number; unit: participants
Arm/Group | HBeAg- at Baseline
Number analyzed (Participants) | 51
participants
  Histological improvement | 21
  No histological change | 17
  Histological worsening | 13

3. Secondary Outcome: Liver Histology Scores in HBeAg Negative Participants With Two Sequential Liver Biopsies During the Period of 104 Weeks
Description: The Knodell/histological activity index (HAI) scoring system that represents the sum of scores for periportal bridging necrosis (0-10: none=0, moderate piecemeal necrosis plus bridging necrosis=5, multilobular necrosis=10); interlobular degeneration and focal necrosis (0-4: none=0, marked=4); portal inflammation (0-4: none=0, marked=4) and fibrosis (0-4: none=0, fibrous portal expansion=1, bridging fibrosis=3, cirrhosis=4) was carried out by two independent pathologists in the HBeAg negative participants with 2 sequential liver biopsies during the period of 104 weeks.
Time Frame: Baseline to Week 104
Population: HBeAg negative chronic hepatitis B participants who underwent liver biopsy at Week 48
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | HBeAg- at Baseline
Number analyzed (Participants) | 51
Points on a scale
  Knodell score at baseline | 8.0 (3.8)
  Knodell score at week 104/withdrawal | 5.4 (2.8)
  Necroinflammation score at baseline | 6.3 (3.0)
  Necroinflammation score at week 104/withdrawal | 3.2 (2.0)
  Fibrosis score at baseline | 1.6 (0.9)
  Fibrosis score at week 104/withdrawal | 2.1 (1.2)

4. Secondary Outcome: Change From Baseline in Median Serum HBV DNA Over Time
Description: The HBV DNA level was tested in blood serum by real-time PCR with the LLD as 300 copies/mL at baseline and Weeks 13, 26, 39, 52, 65, 78, 91, and 104 in a central laboratory.
Time Frame: Baseline and Weeks 13, 26, 39, 52, 65, 78, 91, and 104
Population: Intent-to-Treat (ITT) Population: all HBeAg negative participants who actually received the study medication at least once.
Measure: Median (Full Range); unit: log10 copies/mL
Arm/Group | HBeAg- at Baseline
Number analyzed (Participants) | 533
log10 copies/mL
  Serum HBV DNA Reduction at week 13 | -3.2 [-7.0 to 3.4]
  Serum HBV DNA Reduction at week 26 | -3.5 [-7.1 to 1.4]
  Serum HBV DNA Reduction at week 39 | -3.6 [-7.2 to 2.5]
  Serum HBV DNA Reduction at week 52 | -3.6 [-7.2 to 2.4]
  Serum HBV DNA Reduction at week 65 | -3.7 [-7.2 to 2.9]
  Serum HBV DNA Reduction at week 78 | -3.8 [-7.2 to 2.9]
  Serum HBV DNA Reduction at week 91 | -3.7 [-7.2 to 3.2]
  Serum HBV DNA Reduction at week 104 | -3.7 [-7.2 to 2.1]

5. Secondary Outcome: Number of Participants Achieving ALT Normalization at Week 104
Description: Serum alanine aminotransferase (ALT) normalization was defined as a serum ALT level at or below the upper limit of the normal (ULN) range after a baseline value above the ULN, as determined using central laboratory ranges.
Time Frame: Week 104
Population: Intent-to-Treat (ITT) Population: all HBeAg negative participants who actually received the study medication at least once. A total of 435 participants had a baseline ALT value above the ULN.
Measure: Number; unit: participants
Arm/Group | HBeAg- at Baseline
Number analyzed (Participants) | 435
participants
  ALT normalization | 333
  ALT non-normalization | 102

6. Secondary Outcome: Number of Participants Achieving HBsAg Loss and HBsAg Seroconversion at Week 104
Description: HBsAg loss and HBsAg seroconversion (HBsAg loss and HBsAb detected) were assessed for all participants who were HBeAg negative at Weeks 0 and 104. Confirmed HBsAg loss was defined as undetectable HBeAg.
Time Frame: Week 104
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | HBeAg- at Baseline
Number analyzed (Participants) | 533
participants
  HBsAg loss | 1
  HBsAg seroconversion | 0

7. Secondary Outcome: Number of Participants With ADV-associated Resistance at Week 104
Description: Week 104 serum samples from participants who reached a HBV DNA breakthrough were assessed for the development of ADV (Adefovir dipivoxil) mutations (N236T and A181V) in the HBV polymerase. HBV DNA breakthrough was defined as an increase in HBV DNA level by 1 log10 copies/mL or more from the treatment nadir during Weeks 0 to 104.
Time Frame: Week 104
Population: Intent-to-Treat (ITT) Population: all participants who actually received the study medication at least once.
Measure: Number; unit: participants
Arm/Group | 10 mg Adefovir Dipivoxil (ADV)
Number analyzed (Participants) | 533
participants
  HBV DNA breakthrough | 77
  ADV-associated resistance | 9

8. Secondary Outcome: Number of Participants Achieving HBV DNA ≤300 Copies/mL Over Time
Description: as for outcome 1
Time Frame: Weeks 13, 26, 39, 52, 65, 78, 91, and 104
Population: Intent-to-Treat (ITT) Population: all participants who actually received the study medication at least once. Missing data were not included in statistical analysis.
Measure: Number; unit: participants
Arm/Group | HBeAg- at Baseline
Number analyzed (Participants) | 533
participants
  HBV DNA ≤300 cp/mL, Week 13, n=528 | 262
  HBV DNA ≤300 cp/mL, Week 26, n=525 | 350
  HBV DNA ≤300 cp/mL, Week 39, n=523 | 393
  HBV DNA ≤300 cp/mL, Week 52, n=522 | 413
  HBV DNA ≤300 cp/mL, Week 65, n=514 | 415
  HBV DNA ≤300 cp/mL, Week 78, n=513 | 415
  HBV DNA ≤300 cp/mL, Week 91, n=505 | 421
  HBV DNA ≤300 cp/mL, Week 104, n=488 | 403

9. Secondary Outcome: Number of Participants Achieving Complete Response at Week 104
Description: Complete response was defined as an HBV DNA level ≤ 300 copies/mL by the Roche COBAS AMPLICOR HBV MONITOR Test and ALT normalized for two consecutive visits at least 3 months apart.
Time Frame: Week 104
Population: Intent-to-Treat (ITT) Population: all participants who actually received the study medication at least once.
Measure: Number; unit: participants
Groups:
- 10 mg Adefovir Dipivoxil (ADV: 10 mg ADV tablets once daily for 104 weeks
Arm/Group | 10 mg Adefovir Dipivoxil (ADV
Number analyzed (Participants) | 533
participants | 326

10. Secondary Outcome: Time to Protocol-defined Complete Response Over a 104-week Treatment Period
Description: Time to response was defined as the time to participants achieving protocol-defined complete response at week 104 from baseline. Protocol-defined complete response was an HBV DNA level ≤ 300 copies/mL by Roche COBAS AMPLICOR HBV MONITOR Test and ALT normalized for two consecutive visits at least 3 months apart.
Time Frame: Baseline to Week 104
Population: Intent-to-Treat (ITT) Population: all participants who actually received the study medication at least once.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 10 mg Adefovir Dipivoxil (ADV)
Number analyzed (Participants) | 533
days | 301.6 (147.0)

ADVERSE EVENTS:
Arm/Group | 10 mg Adefovir Dipivoxil (ADV)
Serious Adverse Events (participants affected / at risk) | 5
Other Adverse Events (participants affected / at risk) | 38
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | 10 mg Adefovir Dipivoxil (ADV)
Hepatitis B (Infections and infestations) | 1/533
Alanine aminotransferase increased (Investigations) | 1/533
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/533
Neurilemmoma (Nervous system disorders) | 1/533
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1/533
Cerebral hemorrhage (Vascular disorders) | 1/533
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | 10 mg Adefovir Dipivoxil (ADV)
Nasopharyngitis (Infections and infestations) | 38/533

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.